CLINICAL TRIAL: NCT01178684
Title: Study of Epidermal Nerve Fiber Density, Subcutaneous Fat, and Mitochondrial Parameters in Thai HIV-positive Patients on Long-term Stavudine Treatment and in Thai HIV-negative Patients
Brief Title: Epidermal Nerve Fiber Density, Fat and Mitochondrial Parameters in Thai HIV+ Patients on d4T and HIV- Patients
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Assoc.Prof. Jintanat Ananworanich, MD,PhD, SEARCH Research Foundation
Other Study IDs: SEARCH 014
Record Dates: First submitted 2010-06-11; First posted 2010-08-10 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV
Keywords: ENFD; epidermal nerve fiber density; HIV; HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma PBMC Urine CBC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: HIV-pos on d4T with neuropathy
- 2: HIV-pos on d4T without neuropathy
- 3: HIV-neg without peripheral neuropathy
- 4 HIV-pos on d4T with asymtomatic neuropathy

SUMMARY:
This study will provide the range of Epidermal Nerve Fiber Density (ENFD) typically seen in Thai individuals. ENFD values from Thai HIV-negative subjects without neuropathy will be used as appropriate reference norm for Thai HIV-positive subjects. In particular, comparison of ENFD values from Thai HIV-negative subjects with baseline ENFD values in Thai HIV-positive subjects prior to highly active antiretroviral therapy (HAART) will allow examination of the effect of HIV per se on ENFD. ENFD from Thai HIV-positive subjects on long-term d4T (stavudine) with and without neuropathy will also provide reference ENFD values at the extremes of the disease process i.e. extent of ENFD decrease in subjects with d4T-induced symptomatic neuropathy and in subjects completely free of disease despite d4T treatment for comparison with Thai HIV-positive subjects on short-term d4T in SEARCH 003 study.

DETAILED DESCRIPTION:
The range of changes in epidermal nerve fiber density (ENFD), subcutaneous fat, and mitochondrial function induced by stavudine (d4T)-based therapy is currently not known, globally or specifically in the Thai population. This study will evaluate ENFD and subcutaneous fat and peripheral blood mitochondrial parameters in 4 groups of subjects. Group 1 will include Thai HIV-positive subjects on long-term d4T treatment with symptomatic peripheral neuropathy. Group 2 will include Thai HIV-positive subjects on long-term d4T treatment without peripheral neuropathy. Group 3 will include HIV-negative subjects without peripheral neuropathy.Group 4 will include Thai HIV-positive subjects on long-term d4T treatment with asymptomatic peripheral neuropathy. Information gained from Thai HIV-positive subjects on long-term d4T treatment with and without neuropathy in this study will provide range of positive control values for subjects in the SEARCH 003 study and other studies looking at the influence of antiretroviral agents on peripheral nerve, fat, and mitochondria. Information gained from Thai HIV-negative subjects without neuropathy can be used as negative control values for subjects in the SEARCH 003 study and other studies looking at the influence of HIV or other diseases/pathogens on peripheral nerve, fat, and mitochondria.

Hypothesis

1. HIV-positive patients who have been on long-term d4T treatment with symptomatic peripheral neuropathy will have less ENFD, increased lipoatrophy, and altered mitochondrial function than those on long-term d4T treatment with asymptomatic peripheral neuropathy and those on long-term d4T treatment without peripheral neuropathy.
2. HIV-negative patients without peripheral neuropathy will have more ENFD, no lipoatrophy, and better mitochondrial function than HIV-positive patients.

The SEARCH 003 study will assess the extent of deterioration in ENFD induced by short-term (from entry to 24 weeks) d4T use and the degree of improvement following discontinuation of d4T (from week 24 to 72). However the range of changes in ENFD and in other mitochondrial parameters induced by d4T-based therapy in not known, globally or specifically in the Thai population.

This is a cross-sectional study that will enroll 25 HIV-positive subjects on long-term d4T treatment with symptomatic peripheral neuropathy, 25 HIV-positive subjects on long-term d4T treatment without peripheral neuropathy, 50 HIV-negative subjects without peripheral neuropathy and 25 HIV-positive subjects on long-term d4T treatment with asymptomatic peripheral neuropathy for a one-time assessment.

ELIGIBILITY:
Group 1: HIV-positive subjects on long-term d4T with symptomatic peripheral neuropathy

Inclusion Criteria:

* Documented HIV-1 infection
* Age ≥ 18 years old
* Has Thai national identification card
* Subject on d4T treatment with symptoms of neuropathy which developed after start of d4T therapy
* Evidence of symptomatic persistent symptoms of pain, tingling or numbness of lower extremities AND bilateral lower extremity neuropathy on exam at entry.
* Subject understands the study and is able to sign informed consent
* HIV RNA by PCR < 50 copies/mL

Exclusion Criteria:

* Treatment with concomitant medications (other than d4T) or having conditions (e.g. compressive neuropathy, diabetes, vitamin B12 deficiency, excessive alcohol intake meeting substance dependence criteria by DSM-IV, hepatitis C infection) known to cause neuropathy
* History of allergy to any anesthetic medications
* Pregnancy

Group 2 subjects will meet the same criteria described above for group 1 subjects, but will NOT have symptoms OR signs of neuropathy.

Group 3 subjects will meet the same criteria described above for group 1 subjects, but will NOT have symptoms OR signs of neuropathy and will have documented

Group 4 subjects will meet the same criteria described above for group 1 subject, but will have evidence of symptomatic persistent symptoms of pain, tingling or numbness of lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy five HIV-positive patients on long-term d4T treatment (25 with symptomatic peripheral neuropathy, 25 without peripheral neuropathy and 25 with asymptomatic peripheral neuropathy) and 50 HIV-negative subjects without peripheral neuropathy will be recruited from the Thai Red Cross AIDS Research Centre and the Queen Savang Vadhana Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of nerves in the skin | Baseline
  To compare differences in ENFD between the 4 groups
  * group 1: HIV-positive subjects on long-term d4T with symptomatic peripheral neuropathy
  * group 2: HIV-positive subjects on long-term d4T without peripheral neuropathy
  * group 3: HIV-negative subjects without peripheral neuropathy
  * group 4: HIV-positive subjects on long-term d4T with asymptomatic peripheral neuropathy
Condition of lipoatrophy | Baseline
  To compare differences lipoatrophy between the 4 groups
  * group 1: HIV-positive subjects on long-term d4T with symptomatic peripheral neuropathy
  * group 2: HIV-positive subjects on long-term d4T without peripheral neuropathy
  * group 3: HIV-negative subjects without peripheral neuropathy
  * group 4: HIV-positive subjects on long-term d4T with asymptomatic peripheral neuropathy

SECONDARY OUTCOMES:
Mitochondrial parameters | Baseline
Intracellular concentrations of d4T triphosphate | Baseline
HIV DNA in peripheral blood mononuclear cell (PBMC) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Thailand